CLINICAL TRIAL: NCT04409301
Title: Distress in the Pediatric Oncology Setting: Intervention Versus Natural Adaptation - A Multi-Center Study
Brief Title: Distress in the Pediatric Oncology Setting: Intervention Versus Natural Adaptation
Acronym: MSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Family Life Assurance Company (Aflac Inc.) (Unknown)
Responsible Party: Principal Investigator, Tamara Miller, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00116385
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Cancer
Keywords: Behavioral intervention; Medical setting distress
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Hospitals will be randomized to deliver the intervention or to be a control site. Children will be enrolled to ensure equal sized groups of younger (ages 3-6) and older (ages 7-10) children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSAD Intervention (Experimental): Children receiving cancer treatment in a hospital randomized to the My Special Aflac Duck (MSAD) intervention.
  Interventions: Other: My Special Aflac Duck (MSAD)
- Control Group (Active Comparator): Children receiving cancer treatment in a hospital randomized to be a control hospital. Children in the control hospitals will receive the My Special Aflac Duck (MSAD) at the end of the intervention period.
  Interventions: Behavioral: Standard of care control

INTERVENTIONS:
Other: My Special Aflac Duck (MSAD) — The hospital Child Life Specialist or research team member will introduce the child and parent to My Special Aflac Duck MSAD), with instructions on how to use the duck. MSAD is a robotic toy with an associated app. Children can use MSAD for play, exploring feelings, and describing medical procedures. Intervention hospitals are permitted to provide their standard of care from Child Life with the exception of providing stuffed animal-like objects. Data will be recorded by Child Life or research team member on what tools are used outside of the MSAD.
  Arms: MSAD Intervention
Behavioral: Standard of care control — Sites will follow their individual standard of care from Child Life. Data will be recorded by Child Life on what tools are used. After completion of the 3-month survey, patients at hospitals assigned to not initially receive MSAD will each receive a MSAD.
  Arms: Control Group

SUMMARY:
Children with cancer undergo many procedures as part of their treatment, and are often hospitalized or have frequent clinic visits, which can be distressing. Using robots or toys may be promising interventions as they provide elements of distraction therapy to children undergoing stressful and painful medical procedures. The purpose of this study is to see whether the use of a robotic toy called My Special Aflac Duck will reduce distress in children who have been diagnosed with cancer. This multi-center study will involve 20 children, ages 3-10, at each of 8 hospitals and their parent or guardian. There will be a total of 160 participants enrolled nationally.

DETAILED DESCRIPTION:
Annually in the US, over 12,500 children and adolescents are diagnosed with cancer. Youth with cancer undergo numerous procedures, clinic visits, and hospitalizations as part of their treatment and are often hospitalized or frequently come to clinic for procedures and treatment. These events can be distressing and can contribute to a range of negative emotional and/or psychological outcomes. In younger children, coping with distress and anxiety is mediated by their level of cognitive development and affective regulation. Child Life Specialists assist patients and their families during medical experiences by providing individualized educational and emotional support. Distraction techniques, usually performed by Child Life professionals, appear to be better suited to the cognitive abilities of young children, however, the degree to which distraction results in long-term reductions of child distress has not been well-established. Parent(s)/families are also important factors to consider since they are often active in day-to-day care of pediatric cancer patients. Studies have shown that parents have an active role in supporting and training their children during procedures and aiding in interventions and/or during evaluations.

Multisensory toys involving audiovisual, kinesthetic, and tactile senses, requiring a player's active cognitive, motor, and visual skills, have been utilized as an active distraction technique with the potential of reducing pain and anxiety. Robots are promising interventions as they provide elements of distraction to children undergoing stressful and painful medical procedures. In a previous feasibility study completed by the investigative team, results demonstrate high acceptability of My Special Aflac Duck (MSAD) as a device and as a method of distraction for children coping with treatment for pediatric cancer. In addition, the MSAD animatronic device was shown to provide a fun distraction and was used as a tool for expressing feelings for children with cancer in the hospital.

This is a multi-center efficacy trial coordinated through the Aflac Cancer and Blood Disorder Center at Children's Healthcare of Atlanta (CHOA). Hospitals with pediatric oncology departments will be recruited and will be responsible for the enrollment of patients to participate in this study. All participating hospitals will have dedicated Child Life services. Randomized assignment for this trial will be performed at the hospital level. Four hospitals will be assigned to have patients receive the My Special Aflac Duck (MSAD) animatronic device at study initiation and four hospitals will be assigned to not have patients receive MSAD during the study but will receive MSAD at the end of the study.

The study plans to enroll a total of 160 patients and their parent(s)/guardian(s). Within each hospital, 20 families will be recruited; 10 with children aged 3.00-6.99 years and 10 with children aged 7.00-10.99 years.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3.00-10.99 years
* All cancer diagnoses
* English or Spanish speaking (parent and child)

Exclusion Criteria:

* Patients who receive surgery only will be excluded as they will not have follow-up visits at which to complete the questionnaires
* Patients with cognitive or sensory deficits that would impact being able to interact with MSAD and/or complete questionnaires
* Patients who receive chemotherapy entirely inpatient and never have appointments in the outpatient setting

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in Parent Reported Patient Distress with Distress Thermometer | Baseline, Week 1
  The Distress Thermometer instrument asks respondents to indicate how much distress they are experiencing on a scale from 0 to 10 where 0 = no distress and 10 = extreme distress. Parents will report how much medical setting distress that they observe their children experiencing.

SECONDARY OUTCOMES:
Change in Child-Reported Distress with Distress Thermometer | Baseline, Week 1, Month 1, Month 3
  Children will report patient medical setting distress with the Distress Thermometer. The Distress Thermometer instrument asks respondents to indicate how much distress they are experiencing on a scale from 0 to 10 where 0 = no distress and 10 = extreme distress.
Change in Patient Distress with Distress Thermometer as Reported by Child Life Specialists | Baseline, Week 1, Month 1, Month 3
  Child Life Specialists will report patient medical setting distress with the Distress Thermometer. The Distress Thermometer instrument asks respondents to indicate how much distress they are experiencing on a scale from 0 to 10 where 0 = no distress and 10 = extreme distress.
Change in Parent Report of Pediatric Quality of Life Inventory (PedsQL) - Generic Score | Baseline, Week 1, Month 1, Month 3
  Patient quality of life will be assessed with the generic PedsQL as reported by their parents. The parent report surveys for children aged 5-7 and aged 8-12 include 23 items asking about problems the child experienced in the last month. Responses are given on a scale from 0 (never) to 4 (almost always). Responses are reverse scored and linearly transformed to a scale from 0 to 100. The total scale score is the mean of responses, ranging from 0 to 100 where higher scores indicate better quality of life.
Change Parent Reported in PedsQL - Cancer Module Score | Baseline, Week 1, Month 1, Month 3
  Patient quality of life will be assessed with the PedsQL Cancer Module. Parents will complete the parent report assessment corresponding with the age of their child. The instrument for children aged 5-7 has 26 items and the instrument for children ages 8-12 contains 27 items. Responses are given on a scale from 0 (never) to 4 (almost always). Responses are reverse scored and linearly transformed to a scale from 0 to 100. The total scale score is the mean of responses, ranging from 0 to 100 where higher scores indicate better quality of life concerning cancer.
Change in Child Reported PedsQL - Cancer Module Score | Baseline, Week 1, Month 1, Month 3
  Patient quality of life will be assessed with the PedsQL Cancer Module. Children ages 5 and older will complete the child report assessment corresponding with their age. The instrument for children aged 5-7 has 26 items and the instrument for children ages 8-12 contains 27 items. Responses are given on a scale from 0 (never) to 4 (almost always). Responses are reverse scored and linearly transformed to a scale from 0 to 100. The total scale score is the mean of responses, ranging from 0 to 100 where higher scores indicate better quality of life concerning cancer.
Change in Parent Reported Patient-Reported Outcomes Measurement Information System (PROMIS) - Psychological Stress Experiences Score | Baseline, Week 1, Month 1, Month 3
  Patient stress, as reported by parents, will be assessed with the PROMIS Parent Proxy Report for Pediatric Patients, Psychological Stress Experiences survey. This instrument includes 12 items asking about the child's feelings of stress. Responses are given on a scale of 1 to 5 where 1 = never and 5 = always. Total raw scores range from 12 to 60 with higher scores indicating greater experiences of psychological stress. The total raw score can be converted to a standardized T-score with a mean of 50 and a standard deviation of 10. T-scores greater than 50 indicate greater stress.
Change in Child Reported PROMIS - Psychological Stress Experiences Score | Baseline, Week 1, Month 1, Month 3
  Patient stress, as self-reported by children aged 8 and older, will be assessed with the PROMIS Pediatric Psychological Stress Experiences instrument. This instrument includes 19 items with responses given on a scale from 1 (never) to 5 (always). Total raw scores range from 19 to 95 with higher scores indicating greater experiences of psychological stress. The total raw score can be converted to a standardized T-score with a mean of 50 and a standard deviation of 10. T-scores greater than 50 indicate greater stress.
Change in Parent Reported PROMIS - Positive Affect Score | Baseline, Week 1, Month 1, Month 3
  Positive affect, as reported by parents, will be assessed with the PROMIS Positive Affect instrument. This survey contains 15 items for children ages 3-7 and 18 items for children ages 8-12. Responses given on a scale from 1 (not at all or a little bit) to 4 (very much). Total raw scores are standardized to a T-score with a mean of 100 and standard deviation of 15. Standardized scores greater than 100 indicate greater positive affect.
Change in Child Reported PROMIS - Positive Affect Score | Baseline, Week 1, Month 1, Month 3
  Positive affect, as reported by children aged 8 years and older, will be assessed with the PROMIS Positive Affect instrument. This survey contains 9 items for children ages 8-12. Responses given on a scale from 1 (not at all) to 5 (very much). Total raw scores are standardized to a T-score with a mean of 100 and standard deviation of 15. Standardized scores greater than 100 indicate greater positive affect.
Change in Parent Reported PROMIS - Pain Behavior Score | Baseline, Week 1, Month 1, Month 3
  Patient pain, as reported by parents, is assessed with the PROMIS survey for Pain Behavior. This instrument includes 51 items scored on a scale from 1 to 6 where 1 = had no pain and 6 = almost always had pain. Total raw scores range from 51 to 306. The total raw score can be converted to a standardized T-score with a mean of 50 and a standard deviation of 10. T-scores greater than 50 indicate greater pain.
Change in Child Life Specialist Reported Common Terminology Criteria for Adverse Events (CTCAE) - Anxiety | Baseline, Week 1, Month 1, Month 3
  Patient anxiety is assessed by Child Life Specialists with the CTCAE survey for Anxiety. This instrument includes 3 items asking about the child's symptoms of anxiety. Responses are given on a 4-point scale where 1 = no symptoms and 4 = very bad symptoms. Summed scores range from 3 to 12, where higher scores indicate greater anxiety.
Change in Child Life Specialist Reported Common Terminology Criteria for Adverse Events (CTCAE) - Pain | Baseline, Week 1, Month 1, Month 3
  Patient pain is assessed by Child Life Specialists with the CTCAE survey for Pain. This instrument includes 3 items asking about the child's symptoms of pain. Responses are given on a 4-point scale where 1 = no symptoms and 4 = very bad symptoms. Summed scores range from 3 to 12, where higher scores indicate greater pain.
Change in Parent Reported CTCAE - Depression Score | Baseline, Week 1, Month 1, Month 3
  Parent report of their child's depression is assessed with the CTCAE survey for depression. This instrument includes 2 items asking about the child's symptoms of depression. Responses are given on a 4-point scale where 1 = no symptoms and 4 = very bad symptoms. Summed scores range from 2 to 8, where higher scores indicate greater depression.
Change in Child Reported CTCAE - Depression Score | Baseline, Week 1, Month 1, Month 3
  Children ages 8 and older will self-report depression with the CTCAE survey for depression. This instrument includes 2 items asking about the symptoms of depression. Responses are given on a 4-point scale where 1 = no symptoms and 4 = very bad symptoms. Summed scores range from 2 to 8, where higher scores indicate greater depression.
Change in Child Life Specialist Reported CTCAE - Depression Score | Baseline, Week 1, Month 1, Month 3
  Child Life Specialists will use the CTCAE survey for depression to assess depression in their patients. This instrument includes 2 items asking about the symptoms of depression. Responses are given on a 4-point scale where 1 = no symptoms and 4 = very bad symptoms. Summed scores range from 2 to 8, where higher scores indicate greater depression.
Change in Brief Symptom Inventory 18 (BSI-18) Score | Baseline, Week 1, Month 1, Month 3
  Parent self-report of psychological distress is assessed with the BSI-18. The BSI-18 includes 18 items asking respondents to indicate how bothered they are by symptoms, on a scale from 0 (not at all) to 4 (extremely). The Global Severity Index is the sum of all scores and ranges from 0 to 72 where higher values indicate greater distress.
Parent Reported Satisfaction with the MSAD Intervention | Baseline, Week 1, Month 1, Month 3
  Parents will report their satisfaction with the MSAD intervention in the context of psychosocial programming. Parents will be asked to indicate how satisfied they are with the MSAD for improving their child's adaptation to the medical setting since being diagnosed with cancer. Responses are given on a scale from 0 (extremely unsatisfied) to 10 (extremely satisfied).
Child Reported Satisfaction with the MSAD Intervention | Baseline, Week 1, Month 1, Month 3
  Children aged 8 years and older will report their satisfaction with the MSAD on a scale from 0 (extremely unsatisfied) to 10 (extremely satisfied).
Child Life Specialist Reported Satisfaction with the MSAD Intervention | Baseline, Week 1, Month 1, Month 3
  Child Life Specialists will report their satisfaction with the MSAD intervention in the context of psychosocial programming. Child Life Specialists will be asked to indicate how satisfied they are with the MSAD for improving their patient's adaptation to the medical setting since being diagnosed with cancer. Responses are given on a scale from 0 (extremely unsatisfied) to 10 (extremely satisfied).
Parent Reported Patterns of Utilization of the MSAD Intervention | Baseline, Week 1, Month 1, Month 3
  Parents will report on the utilization of the MSAD intervention in the context of psychosocial programming, by indicating how many minutes per day their child engages with the MSAD in the medical setting.
Child Life Specialist Reported Patterns of Utilization of the MSAD Intervention | Baseline, Week 1, Month 1, Month 3
  Child Life Specialists will report on the utilization of the MSAD intervention in the context of psychosocial programming, by indicating how many minutes per day their patient engages with the MSAD in the medical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Miller, MD, MSCE, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - Children's of Alabama, Birmingham, Alabama
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Kansas City, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Richmond, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No